CLINICAL TRIAL: NCT03341741
Title: Combined Dry Powder Tobramycin and Nebulized Colistin Inhalation in CF Patients
Acronym: CotoCFII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Coto V3.0
Record Dates: First submitted 2017-11-03; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Cystic Fibrosis With Pulmonary Manifestations
Keywords: chronic pulmonary infection
MeSH Terms: interventions — Colistin

STUDY DESIGN:
Intervention Model Description: randomized, open label clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tobramycin powder / Colistin (Experimental): TOBI®Podhaler 2 x 112 mg daily for 2 x 28 days (on/off); and Colistin solution 2 x daily 1 Mega continuously for 112 days
  Interventions: Drug: Tobramycin Powder; Drug: Colistin
- Colistin (Active Comparator): Colistin solution 2 x daily 1 Mega continuously for at least 30 days
  Interventions: Drug: Colistin

INTERVENTIONS:
Drug: Tobramycin Powder — TOBI®Podhaler 2 x 112 mg daily for 2 x 28 days (on/off);
  Other Names: TOBI®Podhaler
  Arms: Tobramycin powder / Colistin
Drug: Colistin — Colistin solution 2 x daily 1 Mega continuously
  Other Names: Colistin solution

SUMMARY:
To assess whether the inhalative combination of Tobramycin/Colistin is more effective in reducing Pseudomonas colony forming units (CFUs) and improvement of lung function than Colistin in mono-therapy.

DETAILED DESCRIPTION:
Cystic fibrosis (CF), the most common autosomal recessive disorder in Western countries, is caused by mutations of the cystic fibrosis transmembrane conductance regulator molecule (CFTR) and affects approximately 40.000 patients in Europe. The majority of CF patients develop chronic pulmonary infections with Pseudomonas aeruginosa. These are normally treated with single antibiotics, administered orally, intravenously or inhalatively. Once the infection becomes chronic, eradication of the pathogen is not any more possible due to biofilm formation of the pathogen and increasing resistance. However, inhalative antibiotic combination therapy might be more efficient than single antibiotic therapy in chronically infected CF patients. This notion is supported by previous in vitro and animal studies using Tobramycin/Colistin combination therapy. Importantly, a pilot study in five CF patients who inhaled consecutively Colistin and Tobramycin solutions for 4 week, revealed a decrease of log10 2.52 ± 2.5 cfu of P. aeruginosa in sputum specimens during the course of the treatment compared to baseline values (p=0.027). The treatment was shown to be safe and well tolerated. However, forced expiratory volume in 1 sec (FEV1) did not differ significantly.

Taking advantage of the new development of dry powder inhalation (DPI) antibiotics, specifically TOBI© Podhaler, a larger randomised trial has been performed in which the combined TOBI© Podhaler and Colistin treatment is compared to the monotherapy with Colistin.

ELIGIBILITY:
Inclusion Criteria:

1. Cystic Fibrosis is verified;
2. Patient is 12 years or older;
3. FEV1 is higher than 25% and lower than 100%;
4. The patients' lung is colonised with P. aeruginosa chronically (≥6 months);
5. P. aeruginosa must be sensitive for Tobramycin or Colistin;
6. Pretreated with Colistin >2 months;
7. Last i.v. antibiotic treatment ≥2 weeks;
8. Informed consent is given by patients/legal representatives

Exclusion Criteria:

1. Clinical deterioration is present (exacerbation symptoms);
2. Last Tobramycin inhalation treatment ≤ 2 weeks;
3. Renal dysfunction (creatinine <1.5 fold of normal, glomerular filtration rate (GFR) <80%) at baseline
4. auditoria or vestibular dysfunction, hearing loss
5. Intolerances against Tobramycin, Colistin or Polymyxin B
6. Myasthenia gravis
7. Porphyria
8. Pregnancy and nursing

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03-11 (Actual); Primary Completion 2015-12-19 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Amount of P. aeruginosa in sputum | 30 days
  The primary endpoint will be the difference of P. aeruginosa cfu/ml in sputum with combined therapy with Tobramycin/Colistin compared to colistin mono-therapy. The analysis will be adjusted for baseline values of each cycle and parametric (paired t-Test) or non-parametric (sign test) methods will be used as appropriate.

SECONDARY OUTCOMES:
Course of P.aeruginosa amount in sputum | 112 days
  Course of P. aeruginosa in sputum measured as cfu/ml during the study
Course of forced vital capacity (FVC) absolute amount | 112 days
  Course of FVC absolute in litres during the study
Course of FVC relative amount | 112 days
  Course of FVC relative (percent of expected amount for given body height and gender) during the study
Course of FEV1 absolute amount | 112 days
  Course of FEV1 absolute in litres during the study
Course of FEV1 relative amount | 112 days
  Course of FEV1 relative (percent of expected amount for given body height and gender) during the study
Course of MEF25-75 absolute amount | 112 days
  Course of MEF25-75 absolute in litres during the study
Course of MEF25-75 relative amount | 112 days
  Course of MEF25-75 relative (percent of expected amount for given body height and gender) during the study
Course of proinflammatory cytokine IL1ß amount | 112 days
  Course of proinflammatory cytokine IL1ß amount in sputum [pg/ml] during the study
Course of proinflammatory cytokine IL6 amount | 112 days
  Course of proinflammatory cytokine IL6 amount in sputum [pg/ml] during the study
Course of proinflammatory cytokine IL8 amount | 112 days
  Course of proinflammatory cytokine IL8 amount in sputum [pg/ml] during the study
Course of antiinflammatory cytokine IL10 amount | 112 days
  Course of antiinflammatory cytokine IL10 amount in sputum [pg/ml] during the study
Course of proinflammatory cytokine TNFa amount | 112 days
  Course of proinflammatory cytokine TNFa amount in sputum [pg/ml] during the study
Course of proinflammatory cytokine GM-CSF amount | 112 days
  Course of proinflammatory cytokine GM-CSF amount in sputum [pg/ml] during the study
Course of DNA amount in sputum | 112 days
  Course of DNA amount {pg/ml] in sputum during the study
Course of leukocyte amount in sputum | 112 days
  Course of leukocyte amount [pg/ml] in sputum during the study
Exacerbation | 112 days
  Number of exacerbations during the study
Antibiotics | 112 days
  Use of antibiotics during the study

IPD SHARING:
Plan to Share IPD: No